CLINICAL TRIAL: NCT05911165
Title: Evaluating the Impact of Video-based Surgical Coaching on Obstetrics and Gynecology Residents' Laparoscopic Suturing Skills
Brief Title: Impact of Surgical Coaching on Resident ObGyn Laparoscopic Skills
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 22-836
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Educational Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Resident participants who do not receive video-based surgical coaching
  Interventions: Other: No surgical coaching
- Comparison group (Experimental): Resident participants who do receive video-based surgical coaching
  Interventions: Other: Surgical coaching

INTERVENTIONS:
Other: No surgical coaching — During the twelve-month study period, all participants will have access to an instructional video related to laparoscopic vaginal cuff suturing and the laparoscopic vaginal cuff trainer in order to practice laparoscopic suturing as desired. All participants will keep a log of voluntary practice time on the vaginal cuff trainer. These resources will constitute the control arm of the study
  Arms: Control group
Other: Surgical coaching — Surgical coaching sessions will include 30-60 minute meetings in which the coach-coachee pair reviews recorded laparoscopic suturing practice sessions to examine different aspects of surgical performance.
  Arms: Comparison group

SUMMARY:
Surgical coaching involves the development of a partnership between two surgeons in which one surgeon (coach) guides the other (coachee) in identifying goals, providing feedback and facilitating action planning. Surgical coaching provides an effective means of acquiring new technical and non-technical skills. In this study, the investigators aim to perform a randomized controlled trial to evaluate the impact of a video-based surgical coaching intervention on laparoscopic closure of the vaginal cuff among Obstetrics and Gynecology residents. Obstetrics and Gynecology resident participants will be randomly assigned to the control or intervention groups. Participants will have access to an instructional video related to laparoscopic vaginal cuff suturing and the validated laparoscopic vaginal cuff trainer to practice laparoscopic suturing as desired. The intervention group will receive the same resources as the control group and will also undergo three video-based coaching sessions focused on laparoscopic suturing on the validated laparoscopic vaginal cuff trainer. Our main outcome will consist of participants' change in technical skills of laparoscopic suturing the vaginal cuff, measured by the change in Global Operative Assessment of Laparoscopic Skills Plus score (Vassiliou 2005) from baseline to study completion. Secondary outcomes will include participants' self-reported surgical confidence, operative enjoyment, and plans to incorporate surgery into their career.

DETAILED DESCRIPTION:
During the twelve-month study period, all participants will have access to an instructional video related to laparoscopic vaginal cuff suturing and the laparoscopic vaginal cuff trainer in order to practice laparoscopic suturing as desired. All participants will keep a log of voluntary practice time on the vaginal cuff trainer. These resources will constitute the control arm of the study.

Participants randomized to the surgical coaching arm (coachees) will also receive three video-based coaching sessions over the course of a twelve-month study period focused on laparoscopic suturing. Surgical coaches will include attendings and gynecologic surgery fellows who are comfortable incorporating laparoscopic suturing of the vaginal cuff at the time of hysterectomy into their own practice. The coaches participating in this study will also be listed as investigators. Surgical coaching sessions will include 30-60 minute meetings in which the coach-coachee pair reviews recorded laparoscopic suturing practice sessions to examine different aspects of surgical performance. The coachee will be responsible for providing a video of their own practice of laparoscopic vaginal cuff closure techniques which may occur in a simulation lab utilizing the validated cuff model or in the operating room. At the Cleveland Clinic, all laparoscopic surgeries at Main Campus are recorded and saved on a secure database in the cloud. Surgeries at the regional campuses, including Hillcrest, Fairview, and South Pointe are also saved on a secure tower within the operating room. These videos are taken from the laparoscopic camera and only show the operative field, without any patient identifying information. These videos are stored and commonly used for surgical review, education, and research purposes. Residents will have access to the intraoperative recordings for which they performed laparoscopic suturing. These videos will be utilized for review during the surgical coaching sessions. Additionally, at the beginning of each coaching session, individualized goals will be set by the coachee in order to facilitate discussion during the session. At the end of each session, the coachee will determine a personal action plan for which they will focus until the following coaching session. As part of the surgical coaching method, the goals and action planning are determined by the coachee based on their specific needs, with help of the coach.

All research will take place within the Women's Health Institute. Coaching sessions will be performed in a quiet and private setting where the only participants are the coach/coachee pair.

Comparison:

* Instructional video of laparoscopic vaginal cuff suturing
* Participants will have access to the laparoscopic vaginal cuff trainer in order to practice laparoscopic suturing as desired

ELIGIBILITY:
Inclusion Criteria:

-Cleveland Clinic Ob/Gyn Resident

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Global Operative Assessment Laparoscopic Skills (GOALS-PLUS) | 1-day
  Video-based review of intraoperative vaginal cuff closure performed by the resident utilizing GOALS-Plus on a scale of 0 (worst score) to 40 (best score)

SECONDARY OUTCOMES:
Surgical Confidence | 1-day
  Participant reported confidence in their laparoscopic surgery skills on a 5 point Likert scale of 1 (very unconfident) to 5 (very confident)
Surgical Confidence | 1 day
  Participant reported confidence in their ability to perform laparoscopic cuff closure on a 5 point Likert scale of 1 (very unconfident) to 5 (very confident)
Enjoyment in the operating room | 1 day
  Participant reported enjoyment in the operating room on a 5 point Likert scale of 1 (very much do not enjoy) to 5 (very much enjoy)
Plans to incorporate surgery into career | 1 day
  Participant reported plans to incorporate surgery into their attending practice on a 4 point Likert scale of 1 (no surgery at all) to 4 (primarily surgery)
Amount of tracking months | 1 day
  Participant reported time spent tracking with a gynecologic surgical subspecialty on a 4 point Likert scale of 1(0 months) to 4 (>3 months)
Surgical experience | 1 day
  Participant reported number of times they have performed a laparoscopic vaginal cuff closure on a 4 point Likert scale of 1 (never) to 4 (>10 times)
Time spent watching instructional videos | 1 day
  Participant reported amount of time spent watching instructional videos on a 5 point Likert scale of 1 (no time) to 5 (>5 hours)
Time spent watching personal surgical videos | 1 day
  Participant reported amount of time spent watching personal surgical videos on a 5 point Likert scale of 1 (no time) to 5 (>5 hours)
Time spent practicing on simulation model | 1 day
  Participant reported amount of time spent practicing vaginal cuff closure on the simulation model on a 5 point Likert scale of 1 (no time) to 5 (>5 hours)
Experience undergoing surgical coaching | 1 day
  Participant reported enjoyment as a coachee undergoing surgical coaching (if applicable) on a 5 point Likert scale of 1(very much enjoyed) to 5 (very much did not enjoy)
Experience undergoing surgical coaching | 1 day
  Participant reported helpfulness of surgical coaching for the advancement of their laparoscopic vaginal cuff closure skills on a 5 point Likert scale of 1 (very helpful) to 5 (very unhelpful)
Experience undergoing surgical coaching | 1 day
  Participant reported likelihood of recommending surgical coaching to a colleague on a 5 point Likert scale of 1 (very likely) to 5 (very unlikely)
Sport confidence assessment instrument | 1 day
  Series of questions asking participants to compare their self-confidence to the most confident surgeon they know. Questions are ranked on a 9 point Likert scale of 1 (low) to 9 (high).

CONTACTS AND LOCATIONS:
Overall Officials: Cara King, D.O., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No